CLINICAL TRIAL: NCT06987994
Title: The Effect of Virtual Reality on Fatigue and Functional Capacity in Patients With Multiple Sclerosis
Brief Title: The Effect of Virtual Reality on Fatigue and Functional Capacity in Patients With MS
Acronym: VRMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRMS2025
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis (MS) - Relapsing-remitting; Virtual Reality
Keywords: multiple sclerosis; virtual reality; fatigue; functional capacity; physical therapy
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Experimental): In this group the number of Participants are 15 . The experment by using VR sessions will last 30 minutes per session, 3 times per week for 4 weeks . In addition to the same physiotherapy program used in the control group, this group will receive Virtual Reality (VR) training using a Meta Quest 2 headset . Patients will interact with immersive environments designed to stimulate movement and functional tasks.
  Interventions: Other: Experemental group
- conventional physica ltherapy (Active Comparator): Participants will receive conventional physiotherapy 3 times per week for 4 weeks. The treatment includes:Standing exercises: multidirectional stepping, single- and double-leg stance .Walking exercises: forward, backward, and lateral walking.Weight-shifting exercises: lunges, half-squats, leaning, and reaching,and the participent will be also 15 pateint
  Interventions: Other: control group( physical therapy)

INTERVENTIONS:
Other: control group( physical therapy) — Participants will receive conventional physiotherapy 3 times per week for 4 weeks. The treatment includes:
  Standing exercises: multidirectional stepping, single- and double-leg stance
  Walking exercises: forward, backward, and lateral walking
  Weight-shifting exercises: lunges, half-squats, leaning, and reaching
  Arms: conventional physica ltherapy
Other: Experemental group — In this group the number of Participants are 15 . The experment by using VR sessions will last 30 minutes per session, 3 times per week for 4 weeks . In addition to the same physiotherapy program used in the control group, this group will receive Virtual Reality (VR) training using a Meta Quest 2 headset . Patients will interact with immersive environments designed to stimulate movement and functional tasks.
  Other Names: Virtual Rrality
  Arms: Virtual Reality group

SUMMARY:
This clinical trial aims to evaluate the effectiveness of virtual reality (VR) as a complementary intervention to traditional physical therapy for individuals diagnosed with Multiple Sclerosis (MS). MS is a chronic neurological condition that affects motor and cognitive functions, with fatigue being one of the most common and disabling symptoms. This study will assess whether the use of VR-based applications, in addition to standard physiotherapy, can reduce fatigue and improve functional capacity in individuals with MS.

Participants will be randomly assigned to two groups: one group will receive conventional physiotherapy only, while the other will receive VR-based therapy alongside physiotherapy. The intervention period will last four weeks, and both groups will be evaluated using standardized outcome measures before and after the intervention. These include the Fatigue Severity Scale (FSS), the Timed Up and Go (TUG) test, and the 6-Minute Walk Test (6MWT).

The study is designed to address a gap in current literature, as no prior research has specifically examined the impact of virtual reality on fatigue and functional performance in MS patients. The findings may provide valuable insights into innovative rehabilitation strategies that enhance patient outcomes and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. individuals diagnosed as MS by a physician
2. Expanded Disability Status Scale (EDSS): 2.0-6.5
3. Patient able to walk with or without the use of unilateral support (e.g., a cane)
4. Patient had not experienced a severe exacerbation of symptoms requiring medical intervention in the previous month
5. subjects had to have the cognitive capacity to assure the requisite cognitive ability
6. spasticity up to 2 on Ashworth scale.

Exclusion Criteria:

* 1. cognitive disorders hampering the execution of the exercises/assessment, 2. Ability to maintain monopodalic-standing position for 10 s 3. cardiovascular disorders 4. orthopedic disorders that could negatively affect balance 5. uncorrected visual or auditory impairments 6. pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Score (FSS) | Baseline and after 4 weeks of intervention
  Fatigue will be assessed using the Fatigue Severity Scale (FSS), a validated questionnaire consisting of 9 items scored on a 7-point Likert scale. The scale measures the impact of fatigue on daily functioning and is widely used in MS populations to evaluate changes in perceived fatigue.

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | Baseline and after 4 weeks of intervention
  The Timed Up and Go (TUG) test will be used to assess functional mobility and fall risk. Participants will be timed as they rise from a seated position, walk 3 meters, turn, walk back, and sit down again. The time (in seconds) required to complete the task will be recorded. TUG is a validated measure commonly used in individuals with MS to assess gait and mobility status.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Istanbul, Turkey (Türkiye)